CLINICAL TRIAL: NCT00788463
Title: A Comparison of Beclomethasone Aqueous Spray and Aerosol Delivery Systems in Nasal Polyps
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-06-542
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Nasal Polyps
Keywords: administration, intranasal; aerosol; beclomethasone; QVAR; corticosteroids; nasal polyps; rhinomanometry; Rhinitis Quality of Life Questionnaire; Quality of Life
MeSH Terms: conditions — Nasal Polyps | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerosol (Experimental)
  Interventions: Drug: Intranasal Beclomethasone aerosol
- Spray (Active Comparator)
  Interventions: Drug: Intranasal Beclomethasone spray

INTERVENTIONS:
Drug: Intranasal Beclomethasone aerosol — Beclomethasone aerosol intranasal, 100ug each nostril, twice daily for 6 months.
  Other Names: QVAR
  Arms: Aerosol
Drug: Intranasal Beclomethasone spray — Beclomethasone spray intranasal, 100ug each nostril, twice daily for 6 months.
  Arms: Spray

SUMMARY:
The purpose of this study is to determine if intranasal Beclomethasone delivered by aerosol or spray is more effective in treatment of nasal polyps.

DETAILED DESCRIPTION:
Aqueous and aerosol delivery of intranasal corticosteroids has never been directly compared previously in patients with nasal polyps and it is unknown whether one is superior.

This objective of this study is to compare the efficacy of intranasal beclomethasone by two different delivery systems, aerosol and aqueous spray in patients with nasal polyps. Primary endpoint is the difference in the overall quality of life as measured by the Rhinitis Quality of Life Questionnaire. The secondary endpoint is the change in Nasal Airflow Resistance as measured by rhinomanometry.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* New diagnosis of nasal polyps confirmed by two physicians

Exclusion Criteria:

* Intranasal corticosteroid use within 4 weeks
* Oral corticosteroids use within 4 weeks
* Oral corticosteroid inhalation (ie for treatment of asthma or COPD) of Budesonide >400ug daily, Fluticasone >250ug daily, Beclomethasone >400ug daily
* Contraindication to intranasal corticosteroid
* Inability to give informed consent
* Participation in another clinical trial
* Pregnancy (or not using effective method of contraception) or lactation
* Cystic fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-11-23 (Actual); Primary Completion 2009-03-30 (Actual); Study Completion 2011-11-30 (Actual)

PRIMARY OUTCOMES:
Difference in overall quality of life as measured by the Rhinitis Quality of Life Questionnaire | 0, 1, 3, 6 months

SECONDARY OUTCOMES:
Difference in Nasal Airflow Resistance as measured an anterior rhinomanometry | 0, 1, 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A Mazza, MD, Principal Investigator — Western University, Canada
Locations (1):
- Allergy Clinic, London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] SILCOX LE. The intranasal use of hydrocortisone alcohol. AMA Arch Otolaryngol. 1954 Oct;60(4):431-9. doi: 10.1001/archotol.1954.00720010443005. No abstract available. PMID 13196789
- [Background] SMITH RE. DEXAMETHASONE NASAL AEROSOL IN NASAL POLYPS AND HYPERTROPHIC ALLERGIC RHINITIS: A CLINICAL AND CONTROLLED EVALUATION. Ann Allergy. 1965 Jun;23:273-6. No abstract available. PMID 14308145
- [Background] Taub SJ. Dexamethasone nasal aerosol vs. placebo in the treatment of nasal polyposis. Eye Ear Nose Throat Mon. 1968 Aug;47(8):392-5. No abstract available. PMID 4891434
- [Background] Norman PS, Winkenwerder WL, Agbayani BF, Migeon CJ. Adrenal function during the use of dexamethasone aerosols in the treatment of ragweed hay fever. J Allergy. 1967 Jul;40(1):57-61. doi: 10.1016/0021-8707(67)90060-3. No abstract available. PMID 5230040
- [Background] Mygind N, Hansen I. Beclomethasone dipropionate aerosol effect on the adrenals in normal persons. Acta Allergol. 1973 Sep;28(3):211-8. doi: 10.1111/j.1398-9995.1973.tb01327.x. No abstract available. PMID 4800886
- [Background] Mygind N, Pedersen CB, Prytz S, Sorensen H. Treatment of nasal polyps with intranasal beclomethasone dipropionate aerosol. Clin Allergy. 1975 Jun;5(2):159-64. doi: 10.1111/j.1365-2222.1975.tb01848.x. PMID 1095246
- [Background] Sorensen H, Mygind N, Pedersen CB, Prytz S. Long-term treatment of nasal polyps with beclomethasone dipropionate aerosol. III. Morphological studies and conclusions. Acta Otolaryngol. 1976 Sep-Oct;82(3-4):260-2. doi: 10.3109/00016487609120899. PMID 790892
- [Background] Pedersen CB, Mygind N, Sorensen H, Prytz S. Long-term treatment of nasal polyps with beclomethasone dipropionate aerosol. II. Clinical results. Acta Otolaryngol. 1976 Sep-Oct;82(3-4):256-9. doi: 10.3109/00016487609120898. PMID 790891
- [Background] Mygind N, Sorensen H, Pedersen CB. The nasal mucosa during long-term treatment with beclomethasone dipropionate aerosol. A light-and scanning electron microscopic study of nasal polyps. Acta Otolaryngol. 1978 May-Jun;85(5-6):437-43. PMID 665215
- [Background] Toft A, Wihl JA, Toxman J, Mygind N. Double-blind comparison between beclomethasone dipropionate as aerosol and as powder in patients with nasal polyposis. Clin Allergy. 1982 Jul;12(4):391-401. doi: 10.1111/j.1365-2222.1982.tb02544.x. PMID 7116616
- [Background] Krouse HA, Phung ND, Klaustermeyer WB. Intranasal beclomethasone in severe rhinosinusitis and nasal polyps. Ann Allergy. 1983 Jun;50(6):385-8. PMID 6344703
- [Background] el Naggar M, Kale S, Aldren C, Martin F. Effect of Beconase nasal spray on olfactory function in post-nasal polypectomy patients: a prospective controlled trial. J Laryngol Otol. 1995 Oct;109(10):941-4. doi: 10.1017/s002221510013172x. PMID 7499945
- [Background] Irifune M, Ogino S, Harada T, Abe Y. Topical treatment of nasal polyps with a beclomethasone dipropionate powder preparation. Auris Nasus Larynx. 1999 Jan;26(1):49-55. doi: 10.1016/s0385-8146(98)00062-5. PMID 10077256
- [Background] Vidgren MT, Kublik H. Nasal delivery systems and their effect on deposition and absorption. Adv Drug Deliv Rev. 1998 Jan 5;29(1-2):157-177. doi: 10.1016/s0169-409x(97)00067-7. PMID 10837586
- [Background] Dunn AM, Wilson RS, Baggott PJ. A comparison of beclomethasone dipropionate aqueous nasal spray and beclomethasone dipropionate pressurized nasal spray in the management of seasonal rhinitis. Postgrad Med J. 1984 Jun;60(704):404-6. doi: 10.1136/pgmj.60.704.404. PMID 6379630
- [Background] Sidwell S. A comparison of the efficacy and tolerance of an aqueous beclomethasone dipropionate nasal spray with the conventional pressurized spray. Curr Med Res Opin. 1983;8(9):659-64. doi: 10.1185/03007998309109815. PMID 6667629
- [Background] Harries MG, Anderson PB, Gibson GJ, Hof ZE, Baggott PJ. A comparison of an aqueous and a pressurized nasal spray of beclomethasone dipropionate in the management of seasonal rhinitis. Pharmatherapeutica. 1984;3(9):623-5. PMID 6374683